CLINICAL TRIAL: NCT03981211
Title: Treatment of HOsPitalised Inpatients for Hepatitis C (TOPIC): Strategic Therapeutic Intervention to Enhance Linkage to Care in People Who Inject Drugs
Brief Title: Treatment of HOsPitalised Inpatients for Hepatitis C (TOPIC): Therapeutic Intervention Enhancing Care Linkage in People Who Inject Drugs
Acronym: TOPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VHCRP1902
Record Dates: First submitted 2019-05-31; First posted 2019-06-10 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis C; Liver Inflammation; Liver Cirrhoses
Keywords: people who inject drugs; injecting related infectious diseases
MeSH Terms: conditions — Hepatitis C; Hepatitis | interventions — glecaprevir; pibrentasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: 8 weeks G/P standard therapy (Experimental): 8 weeks treatment of a three fixed-dose combination of glecaprevir/pibrentasvir 100/40 mg tablets administered once daily with food (standard duration therapy).
  Interventions: Drug: Glecaprevir/Pibrentasvir 100 MG-40 MG Oral Tablet
- Cohort B: 4 weeks SOF/G/P shortened therapy (Experimental): 4 weeks treatment of 1 tablet sofosbuvir 400 mg and a three fixed-dose combination of glecaprevir/pibrentasvir 100/40 mg tablets administered once daily with food (shortened duration therapy).
  Interventions: Drug: Glecaprevir/Pibrentasvir 100 MG-40 MG Oral Tablet; Drug: Sofosbuvir 400 MG + Glecaprevir/Pibrentasvir 100 MG-40 MG Oral Tablet

INTERVENTIONS:
Drug: Glecaprevir/Pibrentasvir 100 MG-40 MG Oral Tablet — 8 weeks of 3 x co-formulated tablets of glecaprevir (100mg) and pibrentasvir (40mg) once daily or 4 weeks of 1 tablet sofosbuvir 400 mg and a three fixed-dose combination of glecaprevir/pibrentasvir 100/40 mg tablets administered once daily
Drug: Sofosbuvir 400 MG + Glecaprevir/Pibrentasvir 100 MG-40 MG Oral Tablet — 4 weeks of 1 x sofosbuvir (400mg) tablet and 3 x co-formulated tablets of glecaprevir (100mg) and pibrentasvir (40mg) once daily
  Arms: Cohort B: 4 weeks SOF/G/P shortened therapy

SUMMARY:
This study will evaluate the proportion of patients achieving confirmed SVR12 (undetectable HCV RNA at time point 12 weeks plus post treatment commencement) in patients hospitalised for IRID (injecting related infectious diseases) and commencing inpatient DAA treatment within public hospital services.

DETAILED DESCRIPTION:
This study will be conducted as a Phase IV, multicentre, sequential cohort trial.

60 participants will be enrolled from participating hospital inpatient services. They will be evaluated for eligibility by the use of rapid point-of-care (POC) confirmation of viraemia in people who inject drugs (PWID) hospitalised for IRID. The period of hospitalisation for management of IRID, particularly when prolonged, may represent an ideal opportunity to engage HCV-infected PWID and a potential important strategy for broader HCV elimination.

Eligible patients will be enrolled into one of two treatment cohorts A and B.

A) 30 patients will immediately commence treatment whilst an inpatient of G/P (glecaprevir/pibrentasvir) with continuation of therapy and follow-up in viral hepatitis services post discharge (standard duration therapy).

Following the successful completion of Cohort A, eligible patients will be enrolled into Cohort B.

B) 30 patients will immediately commence treatment whilst an inpatient of 4 weeks of SOF/G/P (sofosbuvir/glecaprevir/pibrentasvir) with continuation of therapy and follow-up in viral hepatitis services post discharge (short duration therapy).

Any patient with recurrent viraemia during follow-up will be genotyped +/- sequenced to exclude re-infection. If relapse is confirmed the patient will be offered re-treatment with standard of care (SOC) salvage therapy based on results of resistance testing.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible to participate in this study.

1. Have voluntarily signed the informed consent form.
2. 18 years of age or older.
3. Injected drugs within the last 6 months
4. Hospitalised with an IRID with an anticipated inpatient stay of > 1 week

   Participants must meet the following additional inclusion criteria to be treated in this study.
5. HCV RNA positive
6. Compensated liver disease
7. Documented non-cirrhotic at enrolment with a qualifying liver FibroScan ≤ 9.5 kpA
8. If co-infection with HIV is documented, the subject must meet the following criteria:

   1. ART naïve with CD4 T cell count >500 cells/mm3; OR
   2. On a stable ART regimen (containing only permissible ART) for >4 weeks prior to screening visit, with CD4 T cell count ≥200 cells/mm3 and a plasma HIV RNA level below the limit of detection.

Exclusion Criteria:

Participants who meet any of the exclusion criteria are not to be enrolled in this study.

1. Inability or unwillingness to provide informed consent or abide by the requirements of the study
2. Actively intoxicated.

   Participants that meet any of the additional exclusion criteria are not to be treated in this study.
3. History of any of the following:

   b. Clinical hepatic compensation (i.e. ascites, encephalopathy or variceal haemorrhage) c. Solid organ transplant d. History of severe, life-threatening or other significant sensitivity to study drugs (glecaprevir/pibrentasvir/sofosbuvir) or any excipients of the study drugs
4. Creatinine clearance (CLcr) < 30 mL/min at screening (Cohort B only)
5. Pregnant or nursing female
6. Decompensated liver disease
7. Use of prohibited concomitant medications
8. Chronic use of systemically administered immunosuppressive agents (e.g. prednisone equivalent > 10 mg/day for >2 weeks)
9. Prior treatment failure with an NS5A based DAA regimen

Patients without an IRID but who fulfill all other criteria and are admitted with an expected duration of stay > 1 week may also be included at discretion of study team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-12 (Actual); Primary Completion 2025-02-12 (Estimated); Study Completion 2025-02-12 (Estimated)

PRIMARY OUTCOMES:
SVR12 outcomes for all total patient population | 12 weeks post completion of commenced treatment
  To evaluate the proportion of patients achieving confirmed SVR12 (undetectable HCV RNA at time point 12 weeks plus post treatment commencement) in patients hospitalised for IRID and commencing inpatient DAA treatment within public hospital services.

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Prince of Wales Hospital, Randwick, New South Wales
  - St Vincent's Hospital Sydney, Sydney, New South Wales
  - Blacktown Mt Druitt Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - St Vincent's Hospital, Melbourne, Victoria